CLINICAL TRIAL: NCT00993278
Title: Effects of the Atkins Diet Versus a Low Fat Diet on Endothelial Function, Lipid Profiles, and Systemic Markers of Inflammation
Brief Title: Effects of the Atkins Diet Versus a Low Fat Diet on Inflammation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Robert C. Atkins Foundation (Other)
Responsible Party: Principal Investigator, Caroline Apovian, Professor of Medicine and Pediatrics, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-27361
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Cardiovascular Health; Obesity
MeSH Terms: conditions — Obesity | interventions — Diet; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-Carbohydrate (Modified Atkins) Diet (Active Comparator)
  Interventions: Dietary Supplement: Low-Carbohydrate (Modified Atkins) Diet
- Low-Fat (Heart Healthy) Diet (Active Comparator)
  Interventions: Dietary Supplement: Low-Fat (Heart Healthy) Diet

INTERVENTIONS:
Dietary Supplement: Low-Carbohydrate (Modified Atkins) Diet — Low-Carbohydrate (Modified Atkins) Diet
  Arms: Low-Carbohydrate (Modified Atkins) Diet
Dietary Supplement: Low-Fat (Heart Healthy) Diet — Low-Fat (Heart Healthy) Diet
  Arms: Low-Fat (Heart Healthy) Diet

SUMMARY:
The purpose of this research is to assess the effects of a low-carbohydrate (modified Atkins) diet versus a low fat (Heart Healthy) diet on cardiovascular health.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effects of a modified Atkins diet (low carbohydrate and low calorie) and a traditional heart healthy diet (low fat and low calorie) on biochemical markers of inflammation and metabolism, anthropometric measurements, vascular studies of endothelial function, adipose tissue composition, and patient compliance and satisfaction over a twelve week period in healthy men and women. Patients will be recruited from the Nutrition and Weight Management Center at Boston Medical Center. Enrolled subjects will be randomly assigned to a reduced calorie diet (either the Atkins diet or a traditional heart healthy diet), and will be counseled by a dietitian and a physician throughout the study period. The patients will have physical exams, labs, vascular studies of endothelial function, and adipose tissue biopsies at baseline and at twelve weeks to assess progress. Participants dietary compliance will be assessed using food journals and 24 hour recall.

The Atkins diet appears to have potential to reverse the epidemic of obesity-linked cardiovascular disease (CVD) in the United States. Obesity is in effect an inflammatory state in which adipose (fat) tissue releases adipokines- small, inflammatory proteins. High adipokine levels in the blood lead to an inflammatory response, ultimately damaging the endothelial cells which line the blood vessels and increases the risk of vascular disease. Ultimately the effects of these two different diets will be analyzed to help determine if a low carbohydrate, low calorie diet is more beneficial than a traditional heart healthy diet (low fat, low calorie) at reducing the systemic inflammatory response by using physical exam measures, inflammatory blood markers, vascular ultrasound studies, and adipose tissue biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* BMI greater than or equal to 30

Exclusion Criteria:

* Currently pregnant or lactating
* Type 2 diabetes
* Use of oral anti-diabetes medications (with exception of Metformin for control of PCOS)
* Presence of known peripheral arterial or cardiovascular disease
* Change in body weight (greater or equal to 3% within the past 3 months)
* Recent use (within the four weeks prior to screening) of weight loss medications including but not limited to phentermine, sibutramine, orlistat, or over the counter weight loss products
* History of an eating disorder or significant disordered eating behaviors such as binging/purging, abuse of laxatives or diuretics
* History of established renal or hepatic disease
* History of prior bariatric surgery
* Subjects who report routine tobacco use
* Subjects on Angiotensin receptor blockers (medications such as but not limited too Adicant, Losartan, Avapro, Diovan, Micardis, Teveten, Candesarten/thiazide, Ibesarten/thiazide, Valsartan/thiazide, Losarten/thiazide, Telmisarten/thiazide, Teveten/thiazide

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Endothelial function via Flow-Mediated Dilation (FMD) | 3 months

SECONDARY OUTCOMES:
Systemic inflammatory markers | 3 months
Body composition via Dual energy x-ray absorptiometry (DXA) | 3 months
Gene expression of adipose tissue | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Caroline M. Apovian, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ogden CL, Carroll MD, McDowell MA, Flegal KM. Obesity among adults in the United States--no statistically significant change since 2003-2004. NCHS Data Brief. 2007 Nov;(1):1-8. PMID 19389313
- [Background] Kershaw EE, Flier JS. Adipose tissue as an endocrine organ. J Clin Endocrinol Metab. 2004 Jun;89(6):2548-56. doi: 10.1210/jc.2004-0395. PMID 15181022
- [Background] Yancy WS Jr, Olsen MK, Guyton JR, Bakst RP, Westman EC. A low-carbohydrate, ketogenic diet versus a low-fat diet to treat obesity and hyperlipidemia: a randomized, controlled trial. Ann Intern Med. 2004 May 18;140(10):769-77. doi: 10.7326/0003-4819-140-10-200405180-00006. PMID 15148063
- [Background] Brehm BJ, Seeley RJ, Daniels SR, D'Alessio DA. A randomized trial comparing a very low carbohydrate diet and a calorie-restricted low fat diet on body weight and cardiovascular risk factors in healthy women. J Clin Endocrinol Metab. 2003 Apr;88(4):1617-23. doi: 10.1210/jc.2002-021480. PMID 12679447
- [Background] Phillips SA, Jurva JW, Syed AQ, Syed AQ, Kulinski JP, Pleuss J, Hoffmann RG, Gutterman DD. Benefit of low-fat over low-carbohydrate diet on endothelial health in obesity. Hypertension. 2008 Feb;51(2):376-82. doi: 10.1161/HYPERTENSIONAHA.107.101824. Epub 2008 Jan 14. PMID 18195164